CLINICAL TRIAL: NCT01772524
Title: A Parallel Group, Double-Blind, Randomized, Placebo Controlled Phase 1b Trial to Evaluate the Safety, Pharmacokinetics, and Efficacy of a Single Dose of ALD403 Administered Intravenously in Patients With Frequent Episodic Migraines
Brief Title: Safety, Efficacy and Pharmacokinetics of ALD403
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alder Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALD403-CLIN-002
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Migraine
Keywords: Migraine Disorders; Phase 1; ALD403
MeSH Terms: conditions — Migraine Disorders | interventions — eptinezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALD403 (Experimental): Single IV Dose on Day 0
  Interventions: Biological: ALD403
- Saline (Placebo Comparator): Single IV infusion on Day 0
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: ALD403
  Arms: ALD403
Drug: Placebo
  Arms: Saline

SUMMARY:
The purpose of this study is to assess the safety, pharmacokinetics and efficacy of a single dose of ALD403 in the prevention of migraine headache in frequent episodic migraineurs for 24 weeks.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of migraine at ≤ 50 years of age (ICHD-II, 2004 Section 1)
* History of migraine ≥ 12 months with

  * ≥ 5 and ≤ 14 migraine days in each 28 day period in the 3 months prior to screening
  * use of acute migraine medications ≤ 14 days per 28 day period and, within those days, ≤ 10 days of triptan use per 28 day period in the 3 months prior to screening and the 28 day period of completion of eDiary prior to randomization
* Women of child-bearing potential and males with partners of child-bearing potential must agree to use adequate contraception (oral or injectable [depot] estrogen, and/or progestogen, or selective estrogen receptor modulator contraceptive therapeutic, intrauterine contraceptive device, or double barrier method [e.g., condom and diaphragm or spermicidal gel]). Non-childbearing potential is defined as post-menopausal for at least 1 year or surgical sterilization or hysterectomy at least 3 months before screening
* Any hormonal therapy (e.g., oral contraceptives, hormone replacement therapy) use is stable and ongoing for at least 3 months prior to screening and during the 28 day period from screening to randomization
* Agree not to post any personal medical data related to the trial or information related to the trial on any website or social media site (e.g., Facebook, Twitter) until the trial has been completed

Exclusion Criteria

* Confounding pain syndromes including fibromyalgia, chronic musculoskeletal (e.g., low back pain), psychiatric conditions, dementia, or major neurological disorders other than migraine that interfere with the participation in the trial
* Diagnosis of complicated migraine, chronic tension-type headache, hypnic headache, hemicrania continua, new daily persistent headache, basilar, hemiplegic, or familial hemiplegic migraine
* Regular use (greater than 7 days) of prophylactic headache medication (any preventive medication or supplement with evidence of efficacy from at least 1 placebo-controlled trial) within 3 months, or onabotulinumtoxin A within 6 months prior to screening or during the 28 day period prior to randomization
* Cardiac surgery or cardiac symptoms within 3 months of screening and during the 28 day period prior to randomization
* Suspected or diagnosis of hypertension with or without antihypertensive treatment
* Any ongoing co-morbidity that in the opinion of the Investigator will interfere with the participation in the trial
* Body Mass Index (BMI) > 39 at screening
* Pregnant, breast-feeding, or planning to become pregnant during the trial
* Patients who have used opioids > 5 days for the treatment of pain in more than 2 of the 6 months prior to screening or in the 28 day period prior to randomization

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 163 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Safety of ALD403: laboratory variables, ECG and adverse events | 24 weeks
  * Physical Examination
  * Vital signs
  * 12-lead ECG (electrocardiogram)
  * Clinical laboratory tests (hematology, chemistry)
  * Number of participants with Adverse Events

SECONDARY OUTCOMES:
Evaluation of Pharmacokinetics of ALD403 | 24 weeks
  * Cmax - maximum plasma concentration
  * Tmax - Time to achieve maximum plasma concentration
  * AUC - Area under the plasma concentration-time curve
  * T1/2 - Elimination half-life
  * Vz - Volume of distribution
  * CL - Clearance
  * Bioavailability
  * Plasma levels of unbound ALD403
Efficacy of ALD403 | 12 weeks
  * Change in frequency of migraine days compared to baseline
  * Responder rate
  * Migraine hours
  * Migraine episodes
  * Migraine severity
  * Use of acute migraine medications

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Smith, MD, Study Director — Alder Biopharmaceuticals
Locations (26):
- United States (26):
  - Premiere Research, Phoenix, Arizona
  - ACT Trials, Anaheim, California
  - Collaborative Neuroscience Network, Inc., Long Beach, California
  - Medical Center for Clinical Research, San Diego, California
  - San Francisco Clinical Research, San Francisco, California
  - CA Medical Clinic for Headache, Santa Monica, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - MD Clinical, Hallandale, Florida
  - Miami Research, Miami, Florida
  - Segal Institute for Clinical Research, North Miami, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Boston Clinical Trials, Roslindale, Massachusetts
  - MedVadis Research, Watertown, Massachusetts
  - Michigan Headache & Neurological Institute, Ann Arbor, Michigan
  - Clinvest, Springfield, Missouri
  - SPRI, Brooklyn, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - Wake Research, Raleigh, North Carolina
  - Community Research, Cincinnati, Ohio
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - ClinSearch, Chattanooga, Tennessee
  - Neurology Associates of Arlington, Arlington, Texas
  - Premiere Research, Austin, Texas
  - CRI Lifetree, Salt Lake City, Utah
  - Tidewater Integrated Medical Research, Virginia Beach, Virginia
  - Seattle Women's: Health, Research, Gynecology, Seattle, Washington

REFERENCES:
- [Derived] Smith TR, Spierings ELH, Cady R, Hirman J, Ettrup A, Shen V. Cardiovascular outcomes in adults with migraine treated with eptinezumab for migraine prevention: pooled data from four randomized, double-blind, placebo-controlled studies. J Headache Pain. 2021 Nov 25;22(1):143. doi: 10.1186/s10194-021-01360-1. PMID 34823467
- [Derived] Smith TR, Spierings ELH, Cady R, Hirman J, Schaeffler B, Shen V, Sperling B, Brevig T, Josiassen MK, Brunner E, Honeywell L, Mehta L. Safety and tolerability of eptinezumab in patients with migraine: a pooled analysis of 5 clinical trials. J Headache Pain. 2021 Mar 30;22(1):16. doi: 10.1186/s10194-021-01227-5. PMID 33781209
- [Derived] Dodick DW, Goadsby PJ, Silberstein SD, Lipton RB, Olesen J, Ashina M, Wilks K, Kudrow D, Kroll R, Kohrman B, Bargar R, Hirman J, Smith J; ALD403 study investigators. Safety and efficacy of ALD403, an antibody to calcitonin gene-related peptide, for the prevention of frequent episodic migraine: a randomised, double-blind, placebo-controlled, exploratory phase 2 trial. Lancet Neurol. 2014 Nov;13(11):1100-1107. doi: 10.1016/S1474-4422(14)70209-1. Epub 2014 Oct 5. PMID 25297013